CLINICAL TRIAL: NCT02377817
Title: Modifying Maternal Sleep Position in the Third Trimester of Pregnancy With Positional Therapy: A Randomized Pilot Trial
Brief Title: Halifax PrenaBelt Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allan Kember (Other)
Collaborators: Grand Challenges Canada (Other); Innovative Canadians for Change (Other); Global Innovations for Reproductive Health and Life (Other); Kaishin Chu Design (Industry); Nova Scotia Health Authority (Other); University of Michigan (Other); Harvard University (Other)
Responsible Party: Sponsor-Investigator, Allan Kember, Medical Student, IWK Health Centre
Organization: IWK Health Centre (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GCC-S7-0629-01-10-HAL
Record Dates: First submitted 2015-02-17; First posted 2015-03-04 (Estimated); Results first posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Sleep; Pregnancy; Stillbirth; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Very Low Birth Weight; Fetal Growth Retardation; Fetal Hypoxia
Keywords: positional therapy; tennis ball technique; sleep in pregnancy; supine; polysomnography; sleep position; supine position
MeSH Terms: conditions — Stillbirth; Fetal Growth Retardation; Fetal Hypoxia; Deception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PrenaBelt on First Sleep Test Night (Experimental): Participants will be randomized to treatment order: sham PrenaBelt on first night, then PrenaBelt on second night, or vice versa. This will avoid the potential impact of changes to sleep across the two nights resulting from familiarization with the polysomnography equipment, which could bias the results.
  Interventions: Device: PrenaBelt; Device: Sham PrenaBelt
- Sham PrenaBelt on First Sleep Test Night (Sham Comparator): Participants will be randomized to treatment order: sham PrenaBelt on first night, then PrenaBelt on second night, or vice versa. This will avoid the potential impact of changes to sleep across the two nights resulting from familiarization with the polysomnography equipment, which could bias the results.
  Interventions: Device: PrenaBelt; Device: Sham PrenaBelt

INTERVENTIONS:
Device: PrenaBelt — The PrenaBelt is a belt-like, positional therapy (PT) device designed specifically for pregnant women. While the PrenaBelt does not prevent the user from lying on her back or right side during sleep, it is expected to significantly decrease the amount of time she spends in these two positions via the mechanism of PT. PT is a simple, non-invasive, inexpensive, long-established, safe, and effective intervention for preventing people with positional-dependent snoring or obstructive sleep apnea from sleeping on their back - a position that exacerbates their condition.
  The PrenaBelt is worn at the level of the waist. By virtue of its design and position on the user's body, the PrenaBelt affects subtle pressure points on the back and right side of the user when she lies on her back or right side, respectively, activating her body's natural mechanism to spontaneously reposition itself to relieve discomfort, thereby reducing the amount of time she remains on her back or right side.
Device: Sham PrenaBelt — The Sham PrenaBelt and PrenaBelt are the same device except the plastic balls are removed from the Sham PrenaBelt so it cannot provide pressure points.

SUMMARY:
Back and right-sided sleeping position in pregnant women has recently emerged as a potential risk factor for low birthweight (LBW) and stillbirth (SB) in the medical literature. Assuming that sleep position in pregnant women is modifiable, the same literature has indicated that this risk factor is modifiable; however, there is no evidence that this risk factor is truly modifiable.

The proposed link between back and right-sided sleeping position in a pregnant woman and LBW and SB of her baby is multifactorial; however, it ultimately implicates the woman's body position in causing compression of one of the large veins that brings blood back to her heart. This compression, along with other factors relating to the woman, her placenta, and her developing fetus, may result in decreased blood flow (nutrition and oxygen) to her developing baby, which, depending on the extent and duration, could result in LBW or SB of her baby. If the back sleeping position during pregnancy has a causative role in LBW and subsequently SB, the literature indicates that up to 17% of LBW and consequently 26% of SB could potentially be prevented by changing position to avoid back sleep. Note that 20 million LBW and 2.6 million SB occur each year worldwide.

Positional therapy (PT) is a safe and effective intervention for preventing people who snore or people who's breathing pauses during sleep from sleeping on their back - a position that makes their condition worse. The most basic form of PT modifies a person's sleeping position by either:

* Preventing them from sleeping on their back through restricting their movement, or
* Rather than restricting movement, significantly reducing the amount of time they spend sleeping on their back by applying pressure points to their body while they are on their back, which eventually causes them to shift into a different position and avoid lying on their back.

The purpose of this study is to evaluate the ability of a PT intervention to modify the position of pregnant women from their back and right side to their left side while they sleep in late pregnancy.

This study will help determine whether this potential risk factor is modifiable by way of a PT intervention, and whether it is feasible to intervene to reduce or prevent back and right-sided position sleep in late pregnancy. Demonstrating that the sleeping position of pregnant women can be modified through use of a simple, inexpensive PT intervention may be one of the keys to achieving significant reductions in LBW and late SB rates in Canada and worldwide.

DETAILED DESCRIPTION:
The utility of the PrenaBelt in modifying maternal sleeping position and the effect of the PrenaBelt on maternal respiratory and cardiovascular parameters during sleep and sleep staging in the third trimester of pregnancy will be evaluated via a two-night, randomized, cross-over, sham-controlled, triple-blind, sleep study in third trimester pregnant women.

Two nights: one night with a positional therapy (PT) device and one night with sham-PT device to determine treatment effect on outcomes.

Randomized: participants will be randomized to treatment order: sham-PT on first night, then PT on second night, or vice versa. This will avoid the potential impact of changes to sleep across the two nights resulting from familiarization with the equipment, which could bias the results.

Cross-over: on the second night, each participant will be crossed over from PT to sham-PT (or vice versa, depending on randomization order) to allow each participant to act as her own control for comparison of treatment effect on outcomes.

Sham-controlled: a sham-PT device that has the same fit and form of the PT device but without the ability of function (pressure points) will be used as a control. The purpose of a sham-PT device is to identify any specific benefit of one element of a PT device (e.g., fit or form) above and beyond all benefits that might be attributed to everything else about that device (e.g., function). Note that there is no established effective therapy for the population for the indication under study.

Triple blind: participants, sleep technologists monitoring and scoring the sleep tests, and the specialized sleep physician reviewing and reporting the sleep test results will be blinded to the intervention received each night.

Laboratory: conducting this study in a controlled lab setting will allow for continual, real time monitoring of various cardiovascular, respiratory, and sleep parameters of each participant by the sleep technologist. This contributes to a more controlled and safer study overall.

Sleep test: body position, various cardiovascular and respiratory parameters, and sleep parameters will be continuously recorded while the participants are sleeping. Sleep lab procedures will be followed by the personnel conducting, scoring, reviewing, and reporting the sleep tests from participant preparation through discharge

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* low-risk singleton pregnancy
* in the last trimester of pregnancy (≥28 weeks of gestation)
* residing in the Halifax Regional Municipality

Exclusion Criteria:

* BMI ≥ 35 at booking (first antenatal appointment for current pregnancy)
* pregnancy complicated by obstetric complications (hypertension [pre-eclampsia, gestational hypertension, chronic hypertension], diabetes [gestational or not], or intra-uterine growth restriction [<10th %ile for growth])
* sleep complicated by medical conditions (known obstructive sleep apnea, known to get <4 hours of sleep per night due to insomnia, or musculoskeletal disorder that prevents sleeping on a certain side [e.g., arthritic shoulder])
* multiple pregnancy
* known fetal abnormality
* non-English speaking and reading

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2017-01-28 (Actual); Study Completion 2017-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Scott, MD FRCSC, Principal Investigator — The IWK Health Centre
Locations (1):
- IWK Women's Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Owusu JT, Anderson FJ, Coleman J, Oppong S, Seffah JD, Aikins A, O'Brien LM. Association of maternal sleep practices with pre-eclampsia, low birth weight, and stillbirth among Ghanaian women. Int J Gynaecol Obstet. 2013 Jun;121(3):261-5. doi: 10.1016/j.ijgo.2013.01.013. Epub 2013 Mar 15. PMID 23507553
- [Background] Stacey T, Thompson JM, Mitchell EA, Ekeroma AJ, Zuccollo JM, McCowan LM. Association between maternal sleep practices and risk of late stillbirth: a case-control study. BMJ. 2011 Jun 14;342:d3403. doi: 10.1136/bmj.d3403. PMID 21673002
- [Background] Gordon A, Raynes-Greenow C, Bond D, Morris J, Rawlinson W, Jeffery H. Sleep position, fetal growth restriction, and late-pregnancy stillbirth: the Sydney stillbirth study. Obstet Gynecol. 2015 Feb;125(2):347-355. doi: 10.1097/AOG.0000000000000627. PMID 25568999
- [Background] Platts J, Mitchell EA, Stacey T, Martin BL, Roberts D, McCowan L, Heazell AE. The Midland and North of England Stillbirth Study (MiNESS). BMC Pregnancy Childbirth. 2014 May 21;14:171. doi: 10.1186/1471-2393-14-171. PMID 24885461
- [Background] Warland J, Mitchell EA. A triple risk model for unexplained late stillbirth. BMC Pregnancy Childbirth. 2014 Apr 14;14:142. doi: 10.1186/1471-2393-14-142. PMID 24731396
- [Background] O'Brien LM, Warland J. Typical sleep positions in pregnant women. Early Hum Dev. 2014 Jun;90(6):315-7. doi: 10.1016/j.earlhumdev.2014.03.001. Epub 2014 Mar 21. PMID 24661447
- [Derived] Kember AJ, Scott HM, O'Brien LM, Borazjani A, Butler MB, Wells JH, Isaac A, Chu K, Coleman J, Morrison DL. Modifying maternal sleep position in the third trimester of pregnancy with positional therapy: a randomised pilot trial. BMJ Open. 2018 Aug 29;8(8):e020256. doi: 10.1136/bmjopen-2017-020256. PMID 30158217
- See also: Allan Kember's (Project Lead, Project Principal Investigator) blog - Project Updates — https://gojamverandah.wordpress.com/
- See also: Grand Challenges Canada - News Release — https://gojamverandah.files.wordpress.com/2015/01/news-release-grand-challenges-canada-s7-0629-01-10.pdf
- See also: Global Innovations for Reproductive Health and Life — http://www.girhl.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from April 4 2016 through January 27 2017.
  Participants were recruited by a trained nurse a prenatal clinic at the Izaak Walton Killam (IWK) Health Centre, Halifax, Canada, which is a tertiary and primary care center for women and children.
Pre-assignment Details: There was no run-in measurement of baseline sleep habits. The study nights were not required to be consecutive dates. We did not specify a defined washout period. 28 participants were assessed for eligibility. Following exclusion of three who declined participation and two who failed to meet eligibility criteria, 23 were randomized.
Groups:
- PrenaBelt on First Night, Sham PrenaBelt on Second Night: These participants were randomized to receive the PrenaBelt on first night, and the sham-PrenaBelt on second night.
  PrenaBelt: The PrenaBelt is a belt-like, positional therapy (PT) device designed specifically for pregnant women. While the PrenaBelt does not prevent the user from lying on her back or right side during sleep, it is expected to significantly decrease the amount of time she spends in these two positions via the mechanism of PT.
  The PrenaBelt is worn at the level of the waist. By virtue of its design and position on the user's body, the PrenaBelt affects subtle pressure points on the back of the user when she lies on her back, activating her body's natural mechanism to spontaneously reposition itself to relieve discomfort, thereby reducing the amount of time she remains on her back.
  Sham PrenaBelt: The Sham PrenaBelt and PrenaBelt are the same device except the plastic balls are removed from the Sham PrenaBelt so it cannot provide pressure points.
- Sham PrenaBelt on First Night, PrenaBelt on Second Night: These participants were randomized to receive the sham-PrenaBelt on first night, and the PrenaBelt on second night.
  PrenaBelt: The PrenaBelt is a belt-like, positional therapy (PT) device designed specifically for pregnant women. While the PrenaBelt does not prevent the user from lying on her back or right side during sleep, it is expected to significantly decrease the amount of time she spends in these two positions via the mechanism of PT.
  The PrenaBelt is worn at the level of the waist. By virtue of its design and position on the user's body, the PrenaBelt affects subtle pressure points on the back of the user when she lies on her back, activating her body's natural mechanism to spontaneously reposition itself to relieve discomfort, thereby reducing the amount of time she remains on her back.
  Sham PrenaBelt: The Sham PrenaBelt and PrenaBelt are the same device except the plastic balls are removed from the Sham PrenaBelt so it cannot provide pressure points.
Period: Overall Study
Arm/Group | PrenaBelt on First Night, Sham PrenaBelt on Second Night | Sham PrenaBelt on First Night, PrenaBelt on Second Night
Started | 13 | 10
Completed | 10 | 10
Not Completed | 3 | 0
Not completed — Transportation/childcare barriers. | 2 | 0
Not completed — Unrelated injury prevented lateral sleep | 1 | 0

BASELINE CHARACTERISTICS:
Population: Of 23 participants randomized, 3 discontinued participation in the study after the first night, and 20 (10 in each group) completed the study. Baseline demographic, obstetric, and sleep habit characteristics of the 20 participants who completed the study are shown per randomized group (n=10 each).
Groups:
- Total: Total of all reporting groups
Arm/Group | PrenaBelt on First Night, Sham PrenaBelt on Second Night | Sham PrenaBelt on First Night, PrenaBelt on Second Night | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (6.0) | 30.7 (4.1) | 30.9 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 10 | 16
  Filipino | 1 | 0 | 1
  Middle Eastern | 2 | 0 | 2
  Indian | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 10 | 10 | 20
Pre-pregnancy BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.0 (3.3) | 26.2 (3.5) | 26.6 (3.3)
Current BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.9 (3.7) | 29.9 (3.6) | 30.4 (3.6)
Gestational age [Mean (Standard Deviation); unit: weeks] | 30.9 (3.0) | 30.8 (2.8) | 30.9 (2.8)
Gravidity [Count of Participants; unit: Participants]
  Gravida 1 | 4 | 6 | 10
  Gravida ≥2 | 6 | 4 | 10
Nightly sleep duration [Median (Inter-Quartile Range); unit: hours] | 8.0 [7.5 to 8.0] | 7.8 [7.0 to 8.0] | 8.0 [7.0 to 8.0]
In the last week, sleep onset position [Count of Participants; unit: Participants]
  Left | 7 | 10 | 17
  Supine | 3 | 2 | 5
  Right | 8 | 3 | 11
  Prone | 1 | 0 | 1
In the last week, waking position [Count of Participants; unit: Participants]
  Left | 8 | 4 | 12
  Supine | 4 | 4 | 8
  Right | 5 | 6 | 11
  Prone | 0 | 0 | 0
When not pregnant, sleep onset position [Count of Participants; unit: Participants]
  Left | 2 | 3 | 5
  Supine | 3 | 3 | 6
  Right | 2 | 4 | 6
  Prone | 7 | 6 | 13
When not pregnant, waking position [Count of Participants; unit: Participants]
  Left | 5 | 4 | 9
  Supine | 4 | 7 | 11
  Right | 5 | 2 | 7
  Prone | 5 | 4 | 9
Snores ≥3 nights per week [Count of Participants; unit: Participants] | 4 | 3 | 7
Sleeps with bed partner [Count of Participants; unit: Participants] | 7 | 10 | 17
Pillow use [Count of Participants; unit: Participants]
  Under head | 9 | 9 | 18
  Between knees | 8 | 6 | 14
  Behind back | 3 | 5 | 8
  Under tummy | 3 | 4 | 7
  Pregnancy pillow | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage (%) of Sleep Time Supine
Description: Proportion of sleeping time spent in the supine position
Time Frame: 1 night (approximately 8 hours)
Population: Twenty (n=20) participants completed the study. Each of these participants spent two nights in the sleep lab - one night wearing the PrenaBelt and one night wearing the sham PrenaBelt. This constitutes 40 nights (20 nights with the PrenaBelt and 20 nights with the sham PrenaBelt).
Measure: Median (Inter-Quartile Range); unit: percentage of sleep time (%)
Groups:
- PrenaBelt Night: On this night, the participants wore the PrenaBelt.
  PrenaBelt: The PrenaBelt is a belt-like, positional therapy (PT) device designed specifically for pregnant women. While the PrenaBelt does not prevent the user from lying on her back or right side during sleep, it is expected to significantly decrease the amount of time she spends in these two positions via the mechanism of PT.
  The PrenaBelt is worn at the level of the waist. By virtue of its design and position on the user's body, the PrenaBelt affects subtle pressure points on the back of the user when she lies on her back, activating her body's natural mechanism to spontaneously reposition itself to relieve discomfort, thereby reducing the amount of time she remains on her back.
- Sham PrenaBelt Night: On this night, the participants wore the sham PrenaBelt.
  Sham PrenaBelt: The Sham PrenaBelt and PrenaBelt are the same device except the plastic balls are removed from the Sham PrenaBelt so it cannot provide pressure points.
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
percentage of sleep time (%) | 3.5 [0.0 to 16.6] | 16.4 [3.5 to 25.3]

2. Secondary Outcome: Total Sleep Time
Description: This is a standard polysomnography measure of the amount of time the participant spent sleeping during the sleep test.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
minutes | 353 [318 to 376] | 350 [318 to 374]

3. Secondary Outcome: Supine Sleep Time
Description: The time (in minutes) spent sleeping in the supine position.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
minutes | 12.3 [0 to 53.5] | 56.8 [12.4 to 79.1]

4. Secondary Outcome: Left-lateral Sleep Time
Description: Time (in minutes) spent sleeping in the left-lateral position.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
minutes | 185.6 (102.5) | 176.1 (95.2)

5. Secondary Outcome: Right-lateral Sleep Time
Description: Time (in minutes) spent sleeping in the right-lateral position.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
minutes | 108.9 (110.1) | 101.9 (100.9)

6. Secondary Outcome: Percentage Sleep Left
Description: Percentage (%) of sleeping time in the left-lateral position.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of sleep time (%)
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
percentage of sleep time (%) | 57.0 (26.9) | 52.2 (27.0)

7. Secondary Outcome: Percentage Sleep Right
Description: Percentage (%) of sleeping time in the right-lateral position.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of sleep time (%)
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
percentage of sleep time (%) | 31.3 (28.8) | 29.3 (27.5)

8. Secondary Outcome: Sleep Latency
Description: This is a standard polysomnography measure of the amount of time (in minutes) that it takes a participant to transition from full wakefulness to sleep.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
minutes | 11.7 [6.7 to 21.9] | 14.5 [7.2 to 26.2]

9. Secondary Outcome: Sleep Efficiency
Description: This is a standard polysomnography measure of the percentage (%) of time the participant was asleep during the sleep test.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of sleep time (%)
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
percentage of sleep time (%) | 81 [76 to 89] | 83 [79 to 88]

10. Secondary Outcome: Total Arousal Index
Description: This is a standard polysomnography measure of the number of times the participant was aroused from a deeper stage of NREM sleep to a lighter stage, or from REM sleep toward wakefulness. This is reported as a 'total arousal index', which is an average of the number of arousals per hour, and is further classified as a spontaneous, periodic leg movement, or respiratory arousal index.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arousals per hour
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
arousals per hour | 11.2 [8.1 to 18.0] | 12.0 [8.5 to 15.6]

11. Secondary Outcome: Spontaneous Arousal Index
Description: This is a standard polysomnography measure of the number of times the participant was spontaneously aroused from a deeper stage of NREM sleep to a lighter stage, or from REM sleep toward wakefulness. This is reported as an 'arousal index', which is an average of the number of arousals per hour.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: arousals per hour
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
arousals per hour | 10.5 (5.8) | 10.3 (5.5)

12. Secondary Outcome: Periodic Limb Movement Arousal Index
Description: This is a standard polysomnography measure of the number of times the participant was aroused from a deeper stage of NREM sleep to a lighter stage, or from REM sleep toward wakefulness due to periodic limb movements (PLMs). This is reported as an 'arousal index', which is an average of the number of arousals per hour.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arousals per hour
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
arousals per hour | 0 [0 to 1.0] | 0.1 [0 to 0.7]

13. Secondary Outcome: Respiratory Arousal Index
Description: This is a standard polysomnography measure of the number of times the participant was aroused from a deeper stage of NREM sleep to a lighter stage, or from REM sleep toward wakefulness due to respiratory events. This is reported as an 'arousal index', which is an average of the number of arousals per hour.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arousals per hour
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
arousals per hour | 0.4 [0 to 1.1] | 0.4 [0 to 1]

14. Secondary Outcome: Percent Stage 1 Sleep
Description: Percent (%) of total sleep time in sleep stage 1.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of sleep time (%)
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
percentage of sleep time (%) | 9.1 (5.2) | 9.6 (6.0)

15. Secondary Outcome: Percent Stage 2 Sleep
Description: Percent (%) of total sleep time in sleep stage 2.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of sleep time (%)
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
percentage of sleep time (%) | 64.5 (7.4) | 61.0 (8.1)

16. Secondary Outcome: Percent Stage 3 Sleep
Description: Percent (%) of total sleep time in sleep stage 3.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of sleep time (%)
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
percentage of sleep time (%) | 10.9 (8.0) | 11.5 (8.8)

17. Secondary Outcome: Percent REM Sleep
Description: Percent (%) of total sleep time in rapid eye movement (REM) sleep
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of sleep time (%)
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
percentage of sleep time (%) | 15.5 (6.4) | 18.0 (4.6)

18. Secondary Outcome: Apnea Hypopnea Index
Description: Apnea hypopnea index (AHI) is a standard polysomnography measure to indicate the severity of sleep apnea. AHI is the average number of apnea and hypopnea events per hour. Will be reported as a total AHI in units of 'events per hour'.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: events per hour
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
events per hour | 0.5 [0 to 1.5] | 0.5 [0 to 1.5]

19. Secondary Outcome: Respiratory Effort-Related Arousal Index
Description: Respiratory Effort-Related Arousal (RERA) index is a standard polysomnography measure to indicate arousals from respiratory effort. Will be reported in units of 'arousals per hour'.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arousals per hour
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
arousals per hour | 0 [0 to 0.1] | 0 [0 to 0.3]

20. Secondary Outcome: Respiratory Disturbance Index (RDI)
Description: This is a standard polysomnography measure. Like the AHI, RDI reports on respiratory events during sleep, but unlike the AHI, it also includes respiratory-effort related arousals (RERAs). RERAs are arousals from sleep that do not technically meet the definitions of apneas or hypopneas, but do disrupt sleep. Will be reported as a total RDI as well as RDI while supine and RDI while non-supine.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: events per hour
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
events per hour
  Total RDI | 0.65 [0 to 1.5] | 0.55 [0.15 to 1.75]
  RDI while supine | 0 [0 to 0] | 0 [0 to 1.2]
  RDI while non-supine | 0.2 [0 to 1.5] | 0.5 [0 to 1.75]

21. Secondary Outcome: Peripheral Blood Oxygen Saturation (SpO2)
Description: SpO2 measured by fingertip pulse oximetry is a standard measure to indicate the oxygen saturation. Mean SpO2, Min SpO2, and Max SpO2 during Rapid Eye Movement (REM), and Non-REM (NREM) states.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of SpO2 (%)
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
percentage of SpO2 (%)
  REM maximum | 98 [98 to 99] | 98.5 [98 to 99]
  REM mean | 96 [94.9 to 96.7] | 96.3 [95.5 to 97.1]
  REM minimum | 92.5 [90.8 to 94] | 92 [89 to 94]
  NREM maximum | 99.0 [98 to 100] | 99.0 [98 to 100]
  NREM mean | 96.1 [95.6 to 96.6] | 96.3 [95.7 to 97.0]
  NREM minimum | 92 [91 to 94] | 92.5 [89 to 94]

22. Secondary Outcome: Number of Participants With Snoring
Description: This is a standard polysomnography measure of the presence of snoring via nasal cannula (pressure transducer) and by objective report of the research assistant (real-time audio feed).
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
Participants | 15 | 11

23. Secondary Outcome: PrenaBelt User Feedback Questionnaire - Satisfaction
Description: Each participant will complete the PrenaBelt User Feedback Questionnaire.
  On a scale of 1 to 10, participant's level of satisfaction with the PrenaBelt. Note:
  1 = extremely dissatisfied 5-6 = acceptable 10 = extremely satisfied
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
units on a scale | 7.5 [6.0 to 8.3] | 7.5 [5.5 to 9.0]

24. Secondary Outcome: PrenaBelt User Feedback Questionnaire - Comfort
Description: Each participant will complete the PrenaBelt User Feedback Questionnaire. On a scale of 1 to 10, participant's level of comfort while wearing and sleeping with the PrenaBelt. Note:
  1 = extremely uncomfortable 5-6 = acceptable 10 = extremely comfortable
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
units on a scale | 9.0 [6.8 to 9.3] | 9 [7.8 to 10]

25. Secondary Outcome: PrenaBelt User Feedback Questionnaire - Intention to Use
Description: Each participant will complete the PrenaBelt User Feedback Questionnaire. On a scale of 1 to 10, participant's intention to use the PrenaBelt during a subsequent pregnancy if it was available to her.
  Note:
  1 = participant would never use it again 5-6 = participant would consider using it again 10 = participant would certainly use it again
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | PrenaBelt Night | Sham PrenaBelt Night
Number analyzed (Participants) | 20 | 20
units on a scale | 8 [5.8 to 8.0] | 7.0 [6.0 to 9.0]

26. Secondary Outcome: Sleep Onset Position
Description: To determine the accuracy of self-reported sleep behaviours against the gold-standard, polysomnography. This is the sleep onset position (left, supine, right) per the participant's self report and is compared with the sleep onset position (left, supine, right) per the polysomnography data.
Time Frame: 1 night (approximately 8 hours)
Population: 20 participants completed the study and each spent 2 nights in the sleep lab (1 night wearing the PrenaBelt and 1 night wearing the sham PrenaBelt), which is 40 nights (40 self-reports and 40 polysomnography reports). The Arms/Groups are combined in this analysis because the treatment order was not expected to affect the accuracy of self-reporting.
Measure: Count of Units; unit: Nights
Units Other Than Participants: Nights
Groups:
- Self-report: To determine the accuracy of self-reported sleep behaviours against the gold-standard, polysomnography. This data is per the participant's self-report, which was elicited from her via the PrenaBelt User Feedback Questionnaire immediately after waking in the morning. On the night previous, participants were not shown the questionnaire nor told specific details about questions she would be asked via the questionnaire in the morning.
- Polysomnography: This data is per the participant's polysomnography recording.
Arm/Group | Self-report | Polysomnography
Number analyzed (Participants) | 20 | 20
Number analyzed (Nights) | 40 | 40
Nights
  Left | 31 | 29
  Supine | 2 | 3
  Right | 7 | 8
  Prone | 0 | 0

27. Secondary Outcome: Waking Position
Description: To determine the accuracy of self-reported sleep behaviours against the gold-standard, polysomnography. This is the participant's waking position (left, supine, right, prone) per the participant's self report and is compared with the waking position (left, supine, right, prone) per the polysomnography data.
Time Frame: 1 night (approximately 8 hours)
Population: as for outcome 26
Measure: Count of Units; unit: Nights
Units Other Than Participants: Nights
Arm/Group | Self-report | Polysomnography
Number analyzed (Participants) | 20 | 20
Number analyzed (Nights) | 40 | 40
Nights
  Left | 28 | 22
  Supine | 0 | 5
  Right | 12 | 13
  Prone | 0 | 0

28. Secondary Outcome: Number of Position Changes
Description: To determine the accuracy of self-reported sleep behaviours against the gold-standard, polysomnography. This is the number of times the participant changed body position (e.g., supine to left side) per the participant's self report and is compared with the number of times the participant changed body position per the polysomnography data.
Time Frame: 1 night (approximately 8 hours)
Population: Only 15 participants completed this question; each of these spent 2 nights in the sleep lab (1 PrenaBelt night and 1 sham PrenaBelt night), which is 30 nights (30 self-reports and 30 polysomnography reports). The Arms/Groups are combined in this analysis because the treatment order was not expected to affect the accuracy of self-reporting.
Measure: Median (Inter-Quartile Range); unit: position changes
Units Other Than Participants: Nights
Arm/Group | Self-report | Polysomnography
Number analyzed (Participants) | 15 | 15
Number analyzed (Nights) | 30 | 30
position changes | 3 [2 to 4] | 6 [3.3 to 10]

29. Secondary Outcome: Percentage of Total Sleep Time in Each Position
Description: To determine the accuracy of self-reported sleep behaviours against the gold-standard, polysomnography. This is the percentage (%) of total sleep time in each position (left, supine, right, prone) per the participant's self report and is compared with the percentage (%) of total sleep time in each position (left, supine, right, prone) per the polysomnography data.
Time Frame: 1 night (approximately 8 hours)
Population: Of 18 participants that answered this question, all except 1 of these participants answered it on both nights, which yields 35 nights (35 self-reports and 35 polysomnography reports). The Arms/Groups are combined in this analysis because the treatment order was not expected to affect the accuracy of self-reporting.
Measure: Mean (Standard Deviation); unit: percentage of sleep time (%)
Units Other Than Participants: Nights
Arm/Group | Self-report | Polysomnography
Number analyzed (Participants) | 18 | 18
Number analyzed (Nights) | 35 | 35
percentage of sleep time (%)
  Left | 59.9 (28.1) | 54.4 (26.4)
  Supine | 7.8 (20.0) | 14.8 (18.7)
  Right | 31.3 (27.3) | 30.8 (28.5)
  Prone | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: Participants completed their polysomnography studies from April 8 2016 through January 27 2017. Each participant that finished the study completed two full nights (7pm to 7am) in the polysomnography laboratory.
Description: Participants were permitted to remove the intervention and/or polysomnography (PSG) equipment at any point if they became uncomfortable. No participants (including the three who did not complete the study) requested to remove the intervention or PSG equipment. There were no known harms related to the interventions or procedures in this study.
Arm/Group | PrenaBelt on First Night, Sham PrenaBelt on Second Night | Sham PrenaBelt on First Night, PrenaBelt on Second Night
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 0/13 | 0/10

LIMITATIONS AND CAVEATS:
Performed in a controlled sleep laboratory setting over two nights; therefore, caution should be taken when extrapolating the results to the home setting and across the third trimester. Due to the small sample, may have been under-powered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-01-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT02377817/SAP_000.pdf
  • Study Protocol (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT02377817/Prot_001.pdf